CLINICAL TRIAL: NCT02673437
Title: An Observational Post-authorization Safety Specialist Cohort Event Monitoring Study (SCEM) to Monitor the Safety and Utilization of Rivaroxaban (XARELTO®) Initiated in Secondary Care for the Prevention of Atherothrombotic Events in Patients Who Have Had Acute Coronary Syndrome in England and Wales
Brief Title: Rivaroxaban ACS Specialist Cohort Event Monitoring Study
Acronym: ROSE ACS
Status: Completed | Type: Observational
Sponsor: Drug Safety Research Unit, Southampton, UK (Other)
Responsible Party: Sponsor
Other Study IDs: ROSE ACS
Record Dates: First submitted 2016-01-25; First posted 2016-02-03 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban group: Patients who have been prescribed rivaroxaban and antiplatelet therapy for the prevention of atherothrombotic events following ACS.
  Interventions: Other: This is a non-interventional study
- Alternative dual antiplatelet therapy: Patients who have been prescribed alternative dual antiplatelet therapy for the secondary prevention of atherothrombotic events following ACS
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
Rivaroxaban is a medicine which reduces the formation of blood clots. Acute coronary syndrome (ACS) comprises a range of disorders, including heart attack and unstable angina, caused by a sudden reduction in blood flow to part of the heart muscle. This study aims to collect information on the use of rivaroxaban and its safety when used by patients for the prevention of atherothrombotic (plaque rupture leading to a blood clot) events following ACS, during the first three months after starting. This study was requested by the European regulatory body (EMA) which is responsible for the use and safety of medicines. It will last for approximately 3 years and is a national study covering the whole of England and Wales. The study aims to recruit 1193 patients who have been prescribed rivaroxaban and antiplatelet therapy and 1193 patients who have been prescribed alternative dual antiplatelet therapy for the secondary prevention of atherothrombotic events following ACS. Each patient will only be monitored for the first 13 weeks after hospital admission for ACS. Patients who choose to take part will complete a consent form. The patient's care team will be asked to complete a baseline questionnaire about the patient at the time the medicine is given and a further questionnaire up to 16 weeks later, specifically asking about the patient's experiences whilst on the medication. If anything unusual is reported during the observation period, the care team may be asked to fill out a followup questionnaire. With the patient's consent, the study team will also inform the patient's General Practitioner (GP) of their participation in the study and will ask the GP to complete an abridged questionnaire from the patient's medical records. The study team will analyse and aggregate the data, carefully protecting patient confidentiality, to classify adverse events of interest, in particular bleeding events.

ELIGIBILITY:
Inclusion criteria:

* Age 18 years or above
* Patients newly prescribed rivaroxaban in any combination with standard oral antiplatelet therapy for the indication of secondary prevention in patients after ACS
* Patients prescribed dual antiplatelet therapy (contextual cohort) for the indication of secondary prevention after ACS
* Patients have provided signed, informed consent

Exclusion criteria:

* Patients prescribed with oral anticoagulants including rivaroxaban within 6 months prior to the index date for any indication
* Patients commenced rivaroxaban between date of market launch (28th October 2014) for the indication of secondary prevention after ACS and study start (18th September 2015)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly prescribed rivaroxaban in any combination with standard oral antiplatelet therapy or current standard antiplatelet combination therapy (at least dual therapy, but not monotherapy) for secondary prevention in patients after ACS
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2015-09; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Cumulative incident risk of major bleeding, overall and stratified by the following bleeding sites: intracranial, gastrointestinal, urogenital. | During 12 weeks after initiation of treatment with rivaroxaban or alternative anticoagulant therapy
  Cumulative incident risk of major bleeding according to the Thrombolysis In Myocardial Infarction (TIMI) classification of non-coronary artery bypass grafting (non-CABG) Related Bleeding, occurring in the 12 week observation period, overall and stratified by the following bleeding sites: intracranial, gastrointestinal, urogenital.The cumulative incidence will be calculated according to the formula:
  Total number of new cases during 12 week observation period x 100 / Population initially at risk If the observed cumulative incidence from this study falls within the range expected as set by the precision limits of cumulative incidence from clinical trial data, then the null hypothesis (of no difference) will not be rejected.
Rate of major bleeding, overall and stratified by the following bleeding sites: intracranial, gastrointestinal, urogenital. | During 12 weeks after initiation of treatment with rivaroxaban or alternative anticoagulant therapy

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Drug Safety Research Unit (for data collation and analysis only), Southampton, Hampshire
  - Drug Safety Research Unit, Southampton, Hampshire